CLINICAL TRIAL: NCT02073851
Title: A Prospective, Single Arm Feasibility Pilot Study to Evaluate the Safety and Performance of the TriGuard™HDH Embolic Deflection Device in Patients Undergoing Transcatheter Aortic Valve Replacement (TAVR)
Brief Title: DEFLECT II: A Study to Evaluate the Safety and Performance of the TriGuard™HDH in Patients Undergoing TAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keystone Heart (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEFLECT II
Record Dates: First submitted 2014-01-27; First posted 2014-02-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TriGuard™HDH (Experimental): Patients undergoing TAVR will be treated wIth experimental device TriGuard™HDH
  Interventions: Device: TriGuard™HDH

INTERVENTIONS:
Device: TriGuard™HDH — TriGuard™HDH Embolic Deflection Device in patients undergoing Transcatheter Aortic Valve Replacement (TAVR)

SUMMARY:
Pilot study enrolling up to 12 patients at a single investigational site in the Netherlands. Patients for TAVR will be enrolled to receive the Embolic Deflection Device throughout the duration of the TAVR procedure.

DETAILED DESCRIPTION:
Prospective, single center, single arm pilot study enrolling up to 12 patients at a single investigational site in the netherlands. Patients meeting eligibility criteria for TAVR and none of the exclusion criteria will be enrolled to receive the Embolic Deflection Device throughout the duration of the TAVR procedure.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥ 18 years of age.
2. The patient meets indications for transcatheter aortic valve replacement procedure.
3. The patient is willing to comply with specified follow-up evaluations.
4. The patient, or legally authorized representative, has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent, approved by the appropriate Medical Ethics Committee (EC).

Exclusion Criteria:

1. Patients undergoing transcatheter aortic valve replacement via the trans-axillary, subclavian, or direct aortic route
2. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to index procedure per site standard test.
3. Patients with known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure (according to definition) or AMI > 72 hours preceding the index procedure and creatine kinase and creatine kinase fraction have not returned to normal limits at the time of procedure.
4. Patients who are currently experiencing clinical symptoms consistent with new onset AMI, such as nitrate-unresponsive prolonged chest pain.
5. Patients with impaired renal function (estimated Glomerular Filtration Rate [Estimated Glomerular Filtration Rate] <30, calculated from serum creatinine by the Cockcroft-Gault formula).
6. Patients with torturous/unsuitable anatomy as related to major cerebral arteries in the aortic arch that may interfere with device deployment or remain deployed.
7. Patients with a platelet count <100.000 cells/mm³ or >700.000 cells/mm³ or a white blood cell <3000 cells/mm³ within 7 days prior to index procedure.
8. Patients with a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated, or will refuse transfusion.
9. Patients who have received any organ transplant or are on a waiting list for any organ transplant.
10. Poor fluoroscopic visualization due to obesity or other medical reason
11. Hypotension requiring iv/ia medication or other therapy such as resuscitation and defibrillation
12. Patients with known other medical illness or known history of substance abuse that may cause non-compliance with the protocol, confound the data interpretation or is associated with a life expectancy of less than one year.
13. Patients with a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, nitinol, stainless steel alloy, latex, and/or contrast sensitivity that cannot be adequately pre-medicated.
14. Patients with a history of a stroke or transient ischemic attack (TIA) within the prior 6 months.
15. Patients with an active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months.
16. Patients presenting with cardiogenic shock.
17. Patients with severe peripheral arterial disease that precludes the delivery sheath vascular access.
18. Patients with severe calcification/atheroma, friable or mobile atherosclerotic plaque in the aortic arch
19. Patients with contraindication to cerebral MRI.
20. Patients going through unprotected (cerebral embolization) cardiovascular procedure prior, during or post transcatheter aortic valve replacement procedure, before the post-procedure diffusion-weighted magnetic resonance imaging evaluation
21. Patients who have a planned treatment with any other investigational device or procedure during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Device performance | During TAVR procedure
  Device performance will be evaluated for the following functions: Access the aortic arch, Deploy the TriGuard™HDH from the delivery catheter, Position the TriGuard™HDH to cover the cerebral/carotid vessels, Retrieve the TriGuard™HDH system intact

SECONDARY OUTCOMES:
Number of new cerebral lesions | one week post procedure
  The number of new cerebral lesions by diffusion-weighted MRI one week post procedure
Volume of new cerebral lesions | One week post procedure
  The volume of new cerebral lesions by diffusion weighted MRI one week post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Stella, Md., Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands